CLINICAL TRIAL: NCT02295163
Title: Short-term Efficacy of Stellate Ganglion Block in Men to Reduce Hot Flushes Related to Androgen Deprivation Therapy
Brief Title: Stellate Ganglion Block for Hot Flushes in Men Treated With ADT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no participants
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Principal Investigator, Jan Willem Kallewaard phd, Principal Investigator, Rijnstate Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL46979.091.13
Record Dates: First submitted 2014-11-11; First posted 2014-11-20 (Estimated); Last update posted 2021-03-10 (Actual); Status verified 2020-03

CONDITIONS: Prostate Cancer
Keywords: Stellate ganglion block; hot flushes; androgen deprivation therapy; prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms; Hot Flashes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham procedure (Sham Comparator): injection of NACL 0,9% in the stellate ganglion
  Interventions: Procedure: Sham procedure
- Stellate ganglion block (Experimental): injection of Bupivacaine 0,5% in the stellate ganglion
  Interventions: Procedure: Stellate ganglion block

INTERVENTIONS:
Procedure: Stellate ganglion block — 7 ml of 0.5% bupivacaine will subsequently be injected next to the stellate ganglion to produce a sympathetic block.
  Arms: Stellate ganglion block
Procedure: Sham procedure — 7 ml of 0.9 % sodium chloride will subsequently be injected next to the stellate ganglion
  Arms: Sham procedure

SUMMARY:
Androgen deprivation therapy (ADT) is widely used as standard therapy in the treatment of locally advanced and metastatic prostate cancer. Hot flushes and night sweats are one of the main side-effects of ADT. There are no successful and well-tolerable treatment options available. A possible treatment for hot flushes is stellate-ganglion block (SGB), used as a means of interrupting parts of the sympathetic nervous system involved in temperature regulation.

Objective of this study:

To assess the short-term efficacy of stellate ganglion block on hot flush reduction versus sham procedure

DETAILED DESCRIPTION:
Androgen deprivation therapy (ADT) is widely used as standard therapy in the treatment of locally advanced and metastatic prostate cancer. Hot flushes and night sweats are one of the main side-effects of ADT. There are no successful and well-tolerable treatment options available. A possible treatment for hot flushes is stellate-ganglion block (SGB), used as a means of interrupting parts of the sympathetic nervous system involved in temperature regulation.

Objective of this study

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age: >18 years
* Mean daily flush frequency of 10 or more and a hot flush score of 15 or more
* Treatment with ADT because of prostate cancer
* Absence of any other cause of flushing

Exclusion Criteria:

* Use of medication that affects flushing: oestrogens, progestogens, clonidine, naloxone, paroxetine, fluoxetine, venlafaxine, gabapentin, luteinizing hormone-releasing hormone receptor antagonist
* Still receiving chemotherapy of radiotherapy
* Psychiatric disease
* Any unstable concurrent disease
* Allergic reactions against bupivacaine or contrast media.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2021-01 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Hot flush score | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: jw. kallewaard, MD, Principal Investigator — Rijnstate Hospital
Locations (1):
- Rijnstate Hospital, Arnhem, Gelderland, Netherlands